CLINICAL TRIAL: NCT02171676
Title: A Phase I Open-label Dose Escalation Study of Single Oral Daily Doses of BIBW 2992 for Three Days After Administration of Docetaxel, in Patients With Advanced Solid Tumors
Brief Title: BIBW 2992 After Administration of Docetaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.20
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel; Afatinib

ARMS (1):
- Docetaxel + BIBW 2992 (Experimental): Dose escalation
  Interventions: Drug: Docetaxel; Drug: BIBW 2992

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere
Drug: BIBW 2992

SUMMARY:
Maximum tolerated dose (MTD), safety, pharmacokinetic and pharmacodynamic parameters, and efficacy of pulsatile administration of BIBW 2992 in combination with docetaxel (Taxotere®)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumors, of types historically known to express EGFR and/or HER2, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment preferably patients with breast, prostate, or ovarian cancer. In addition, patients with a disease amenable for standard treatment with docetaxel
* Age 18 years or older
* Life expectancy of at least three (3) months
* Written informed consent that is consistent with International Conference on Harmonization - Good Clinical Practice guidelines
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
* Patients recovered (Common Terminology Criteria (CTC) Grade 0 or 1) from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies
* Patients recovered from previous surgery

The 12 additional patients recruited at the MTD must also meet the following criteria:

* Measurable tumor deposits (Response Evaluation Criteria in Solid Tumors) by one or more techniques (X-ray, CT, MRI) and/or recognized tumor markers such as prostate specific antigen (prostate cancer) or cancer antigen 125 (Ovarian cancer)

Exclusion Criteria:

* Active infectious disease
* Gastrointestinal disorders that might interfere with the absorption of the study drug or chronic diarrhea
* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
* Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least eight weeks, no history of cerebral edema or bleeding in the past eight weeks and no requirement for steroids or anti-epileptic therapy
* Cardiac left ventricular function with resting ejection fraction CTC ≥ Grade 1
* Absolute neutrophil count (ANC) less than 1500 / mm3
* Platelet count less than 100 000 / mm3
* Bilirubin > upper limit of normal (ULN)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) > 1.5 x ULN
* Alkaline Phosphatase > 2.5 x ULN
* Serum creatinine > 1.5 mg / dl (> 132 μmol / L, SI (Système Internationale) unit equivalent)
* Women and men sexually active and unwilling to use a medically acceptable method of contraception
* Pregnancy or breast-feeding
* Treatment with other investigational drugs; chemotherapy, immunotherapy, radiotherapy or hormone therapy (excluding luteinising hormone-releasing hormone agonists, other hormones taken for breast cancer, or bisphosphonates) or participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
* Treatment with an EGFR- or HER2 inhibiting drug within the past four weeks before start of therapy or concomitantly with this study (8 weeks for trastuzumab)
* Patients unable to comply with the protocol
* Active alcohol or drug abuse
* Hypersensitivity to docetaxel or any component or other drug formulated with polysorbate 80

The patient may be eligible for re-treatment after the previous course is finished. The patient will not be eligible if any of the following conditions are met:

* If patients latest X-ray, CT or MRI reveals progressive disease, or if clinical assessment reveals signs of disease progression
* Cardiac left ventricular function CTC Grade ≥ 2 at any time during the previous course
* Patients fulfilling any of the Exclusion Criteria listed before as determined on day 18 of the treatment course 1 (visit 7) or day 18 (visit R5) of the previous course
* Patients not recovered from any dose-limiting toxicity (DLT) 14 days after onset. Recovery is defined as a return to baseline level or CTC Grade <= 1, whichever is higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 168 days
Incidence and intensity of adverse events according to Common Terminology Criteria for Adverse Events (CTCAE version 3.0) | up to 35 months

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) for different time points | up to 48 hours after the first drug administration
Percentage of AUC0-∞ that is obtained by extrapolation (%AUC0-tz) | up to 48 hours after the first drug administration
Pre-dose plasma concentration (Cpre) | pre-dose on day 3 and 4
Plasma concentration at 24 h following the first (C24,1) dose | 24 hours after the first drug administration
Maximum measured plasma concentration (Cmax) | up to 48 hours after the first drug administration
Time from dosing to the maximum plasma concentration following the first dose of uniform intervals τ (tmax) | up to 48 hours after the first drug administration
Terminal rate constant in plasma (λz ) | up to 48 hours after the first drug administration
Terminal half-life (t1/2) | up to 48 hours after the first drug administration
Mean residence time after oral administration (MRTpo) | up to 48 hours after the first drug administration
Apparent clearance (CL/F) | up to 48 hours after the first drug administration
Apparent volume of distribution (V) for different time points | up to 48 hours after the first drug administration
Modulation of biomarkers (EGFR (Epidermal growth factor receptor), p-EGFR, p-MAPK (mitogen-activated protein kinase), p-Akt, Ki 67, p27Kip1) in skin biopsies | Baseline and day 4
Modulation of biomarkers (EGFR, p-EGFR, HER2 (Human epidermal growth factor receptor), p-MAPK, p-Akt, Ki 67, p27Kip1) in tumour biopsies in 6 or more patients treated at the MTD | Baseline and day 4
Objective tumor response | up to 35 months
Correlation of EGFR, HER2, estrogen receptor (ER) and progesterone receptor (PrR) immunohistochemical status as based on tumor biopsies, or excisions obtained prior to this trial, with objective tumor responses | up to 35 months